CLINICAL TRIAL: NCT06240117
Title: Impact of Intraoperative Cell Salvage on Maternal Hemoglobin, Need for Allogeneic Blood Transfusion and Recovery Time in Women Presenting With Preoperative Moderate Anemia Undergoing Elective Cesarian Section
Brief Title: Impact of Intraoperative Cell Salvage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Under enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-01380
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Peripartum Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care with intraoperative cell salvage (Experimental): Participants for elective surgery with anemia randomized to standard of care with intraoperative cell salvage.
  Interventions: Procedure: Intraoperative cellular salvage
- Standard of care without intraoperative cell salvage (No Intervention): Standard of care for cesarean sections as per the policy of the anesthesiology department.

INTERVENTIONS:
Procedure: Intraoperative cellular salvage — When the patient is randomized to this intervention the cell salvage machine will be set up for intraoperative use. The surgical team will collect blood from the surgical field into the cell salvage machine, which will process the blood for reinfusion. The volume of blood available for reinfusion is determined by the amount of blood lost which can be collected into the cell salvage system. The blood collected into the salvage system will be collected and processed per standard operating room procedure. At least 100mL of blood collected in the system are necessary for processing. If >100mLs are collected, they will be processed and reinfused. The need for additional blood products and medications will be determined by the anesthesiology team based on the patient's hemodynamic status and will proceed per standard of care.
  Arms: Standard of care with intraoperative cell salvage

SUMMARY:
Patients presenting for elective cesarean section will be screened for pre-procedural anemia. If the potential subject meets the selection criteria they will be presented with the option of participating in the study. Once consented the participant is randomized by envelope. The two groups studied are: standard of care with intraoperative cell salvage and standard of care without cell salvage. If the participant is randomized to the cell salvage group, the study team will notify the anesthesia and obstetrics (OB) team and will set up the cell salvage system per protocol. The primary end point is to determine the difference in postoperative hemoglobin at 48hrs, need and quantity of allogeneic blood product transfusion, length of hospital stay between the two groups studied. The secondary endpoints Investigate the impact of using IOCS on clinical parameters associated with maternal postpartum stability and well being and include estimation of blood loss, need for pressors, uterotonics, return to the operating room, uterine compression devices, ICU admission, postoperative blood product transfusion, IV iron supplementation, blood chemistry, coagulation parameters, oliguria, diagnosis of acute kidney injury, postoperative dialysis, acute respiratory distress syndrome, pulmonary edema, pneumonia, deep vein thrombosis, pulmonary embolism, oxygen requirement, new arrythmias APGAR scores, anemia fatigue scale at 24hr and 48 hrs, OBSQOR10 score 24 hours and 48 hours postpartum and 6 week postpartum EPDS score.

ELIGIBILITY:
Inclusion criteria:

* Women aged 18-55 years.
* Presenting for elective cesarean section.
* With hemoglobin less or equal to 11 mg/dL.
* Able to provide informed written consent.

Exclusion criteria:

* Refusal of blood product administration.
* Refusal of intraoperative blood salvage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
The difference in postoperative hemoglobin at 48hrs compared to preoperative baseline | Baseline and 48 hours postoperatively
  The difference in postoperative hemoglobin at 48hrs
Number of participants requiring allogeneic blood product transfusions | at hospital discharge, likely within 120 hours from admission
  Need of allogeneic blood product transfusions
Quantity of allogeneic blood product transfusion in number of packed red blood cells transfused | at hospital discharge, likely within 120 hours from admission
  Quantity of allogeneic blood product transfusion
Total blood volume transfused | at hospital discharge, likely within 120 hours from admission
  Total blood volume transfused
Length of hospital stay | at hospital discharge, likely within 120 hours from admission
  Length of hospital stay

SECONDARY OUTCOMES:
Quantitative blood loss | within 30 minutes of the end of the surgical procedure (approximately 2 hours)
  The quantitative blood loss is obtained from the measured blood lost and accumulated into the measuring devices such as suction canisters and cell saver machine available in the operating room.
Number of participants being administered uterotonics | within 30 minutes of the end of the surgical procedure (approximately 2 hours)
  Uterotonic use is documented by the anesthesiologist when given intraoperatively. They include oxytocin, misoprostol, methylergonovine and carboprost.
Time to first dosage of pressors | Until hospital discharge, likely within 120 hours from admission
  When low blood pressure is measured postoperatively, pressors may be needed for hemodynamic stability. Possible blood pressors used postoperatively include phenylephrine, ephedrine, norepinephrine and epinephrine. The timing will be recorded.
APGAR Scores | at 1 minute post-delivery
  APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low. APGAR scores will be obtained at 1 minute post-delivery.
APGAR Scores | at 5 minutes post-delivery
  APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low.
  APGAR scores will be obtained at 5 minutes post-delivery.
Anemia-Fatigue Scale (FACIT-F) Score | at 24 hours postpartum
  The anemia-fatigue scale (FACIT-F) is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Each item is measured on a Likert scale which ranges from 1-5. The overall score ranges from 0-160, a higher score indicates greater quality of life.
Anemia-Fatigue Scale (FACIT-F) Score | at 48 hours postpartum
  The anemia-fatigue scale (FACIT-F) is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Each item is measured on a Likert scale which ranges from 1-5. The overall score ranges from 0-160, a higher score indicates greater quality of life.
The Obstetric Quality of Recovery-10 (OBSQOR-10) Score | at 24 hours postpartum
  The Obstetric Quality of Recovery-10 patient-reported outcome measure (OBSQOR-10) at 24 hours postpartum is a validated tool for assessing the quality of postpartum recovery. Consists of 10 questions with a scale that ranges from 1-10.
The Obstetric Quality of Recovery-10 (OBSQOR-10) Score | at 48 hours postpartum
  The Obstetric Quality of Recovery-10 patient-reported outcome measure (OBSQOR-10) at 48 hours postpartum is a validated tool for assessing the quality of postpartum recovery. Consists of 10 questions with a scale that ranges from 1-10.
The Edinburgh Postnatal Depression Scale (EPDS) Score | Up to 6 weeks postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) is a short 10-item self-report questionnaire designed to identify mothers at risk for prenatal and postnatal depression will be performed at 6 weeks postpartum. Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder.
Use of postoperative uterine compression devices | Until hospital discharge, likely within 120 hours from admission
  In cases of postoperative bleeding, uterine compression devices may be needed. The use will be recorded.
Timing of postoperative uterine compression devices | Until hospital discharge, likely within 120 hours from admission
  In cases of postoperative bleeding, uterine compression devices may be needed. The timing will be recorded.
Use of postoperative blood product transfusion | Until hospital discharge, likely within 120 hours from admission
  Blood products may be needed postoperatively depending on patient symptoms and laboratory values. The timing of postoperative blood product transfusion will be recorded in relation to the end of procedure time. Possible blood products include packed red blood cells, platelets, fresh frozen plasma and cryoprecipitate.
Amount of postoperative blood product transfusion | Until hospital discharge, likely within 120 hours from admission
  Blood products may be needed postoperatively depending on patient symptoms and laboratory values. The amount of postoperative blood product transfusion will be recorded. Possible blood products include packed red blood cells, platelets, fresh frozen plasma and cryoprecipitate. Will be reported as number of units.
Number of participants receiving postoperative intravenous iron | Until hospital discharge, likely within 120 hours from admission
  Intravenous iron is used in some cases of postoperative anemia. The number of participants receiving postoperative intravenous iron will be recorded.
Number of participants admitted to intensive care unit (ICU) | Until hospital discharge, likely within 120 hours from admission
  When a higher level of care is needed that which can be provided on the post-operative labor and delivery floor, intensive care unit (ICU) admission may be required. The number of participants requiring ICU admission will be recorded.
The timing for intensive care unit (ICU) | Until hospital discharge, likely within 120 hours from admission
  When a higher level of care is needed that that which can be provided on the post-operative labor and delivery floor, intensive care unit (ICU) admission may be required. The timing for ICU admission will be recorded.
Reason for intensive care unit (ICU) | Until hospital discharge, likely within 120 hours from admission
  When a higher level of care is needed that that which can be provided on the post-operative labor and delivery floor, intensive care unit (ICU) admission may be required. The reason for ICU admission will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be included in the URL field below).